CLINICAL TRIAL: NCT00401219
Title: An Open-Label, Single-Dose, Randomized, 4-Period, Crossover, Bioavailability Study Among 3 New Formulations of Premarin 0.625 mg/Medroxyprogesterone Acetate (Mpa) 2.5 mg Compared With a Reference Formulation of Premarin/Mpa (Prempro) 0.625 mg/2.5 mg in Healthy Postmenopausal Women
Brief Title: Study Comparing Bioavailability of 3 New Formulations of Premarin/MPA With Premarin/MPA (PREMPRO) Reference Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0713E1-136
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-12

CONDITIONS: Estrogen Replacement Therapy
MeSH Terms: interventions — Estrogens, Conjugated (USP); Progestins

INTERVENTIONS:
Drug: conjugated estrogens/progestin (MPA)

SUMMARY:
This study will compare the bioavailabity of three new investigational combination formulations of Premarin and medroxyprogesterone acetate (MPA) with a currently marketed formulation of Premarin and MPA, Prempro™. Prempro™ is indicated for use after menopause in women with a uterus to reduce moderate to severe hot flashes; to treat moderate to severe dryness, itching, and burning, in and around the vagina; and to help reduce your chances of getting osteoporosis (thin weak bones). The purpose of this study is to determine if these new formulations of Premarin/MPA provide the same levels of estrogen and MPA in the blood as Prempro in healthy postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, postmenopausal women ages 35 to 70 years, inclusive.
* Naturally postmenopausal women must not have had a menstrual period for at least six months, but less than 12 months, as confirmed by a blood test; or for at least 12 months with no blood hormone test confirmation. Naturally postmenopausal women must not have had a menstrual period since the age of 54. Surgically menopausal women must have undergone bilateral oophorectomy (removal of both ovaries) at least 6 months prior to the start of the study, and the surgical report may be requested to confirm the surgery date and that the surgery was not due to a cancerous condition.
* Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history. Must be able to abstain from smoking during the inpatient stay.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2006-11; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic blood samples for unconjugated and total (unconjugated plus conjugated) estrogens and MPA will be obtained. The following pharmacokinetic parameters will be determined: Cmax, Tmax, t½, AUC0-T, AUC0-¥.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer